CLINICAL TRIAL: NCT01089595
Title: Open Label Phase II Randomized Trial of Tasigna (Nilotinib) 400 mg Twice Daily Alone or in Combination With Gleevec (Imatinib Mesylate) 400 mg Daily for Patients With Advanced GIST That Have Progressed on High Dose Imatinib
Brief Title: Trial of Tasigna (Nilotinib) 400 mg Twice Daily Alone or With Gleevec (Imatinib Mesylate) 400 mg Daily for Patients With Advanced Gastrointestinal Stromal Tumor (GIST)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis is ending their research program for Nilotinib in GIST.
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-SAR-023
Record Dates: First submitted 2010-01-28; First posted 2010-03-18 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: GIST; Metastatic Disease
Keywords: Imatinib Resistance; GIST; Advanced Disease; Nilotinib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (Active Comparator): Nilotinib 400 mg po bid
  Interventions: Drug: Nilotinib
- Nilotinib + Imatinib (Active Comparator): Nilotinib 400 mg BID with Imatinib 400 mg daily
  Interventions: Drug: Nilotinib with Imatinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 400 mg po bid
  Other Names: Tasigna
  Arms: Nilotinib
Drug: Nilotinib with Imatinib — Nilotinib 400 mg po BID Imatinib 400 mg po daily
  Other Names: Tasigna; Gleevec
  Arms: Nilotinib + Imatinib

SUMMARY:
Patients with advanced GIST are treated with imatinib. This study seeks to look at a new therapeutic agent at the time of tumor progression following treatment with 600-800 mg daily of imatinib. The study is looking to see if Nilotinib (tasigna) alone or in combination with imatinib (gleevec) is more effective at controlling disease.

DETAILED DESCRIPTION:
Resistance to imatinib does develop and represents a major clinical challenge. Mechanisms implicated in imatinib resistance include: target resistance due to new KIT or PDGFRA mutations or over expression of the KIT protein; target modulation due to activation of an alternate receptor tyrosine kinase protein with loss of KIT oncoprotein expression; functional resistance due to KIT or PDGFRA activation without a secondary mutation; and alterations in imatinib uptake by P-glycoprotein.

This study seeks to test nilotinib alone and nilotinib in combination with imatinib in patients that have progressed on imatinib.

Nilotinib is a new synthetic second-generation inhibitor of the BCR-ABL tyrosine kinase that competes for the ATP-bindings sites of BCR-ABL. A completed phase I trial assessed the activity of nilotinib alone and in combination with imatinib in patients that have progressed on imatinib in a population of patients with imatinib refractory and intolerant patients. There were rare responses, but stable disease was observed in grater than 50% of patients.

This study is aiming to treat patients with advanced or metastatic GIST who have disease progression on imatinib dose escalated up to 600 mg or greater. The rationale for exploring Nilotinib in this setting is to determine if it has therapeutic efficacy, with potentially less toxicity than the current standard of care for second line therapy. In addition, since it is not uncommon to see progression of some metastatic GIST lesions on imatinib, while others remain controlled, adding nilotinib may treat the progressing lesions while imatinib continues to control the areas without disease progression.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed GIST.
* advanced/metastatic GIST.
* experienced failure of prior treatment with imatinib 600-800 mg per day defined by progression of disease according to RECIST criteria during treatment. Radiographic evidence of PD on imatinib must be confirmed by the Investigator prior to enrollment.
* May have focal progression of disease including a new enhancing nodular focus within a pre-existing tumor nodule; such a nodule should be considered measurable by standard RECIST criteria.
* measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* At least 4 weeks since prior therapy with imatinib & resolution of all acute toxic effects of the prior therapy or surgical procedure to grade ≤1.
* Age >18 years.
* ECOG performance status 0-2.
* Normal organ and marrow function as defined below:

  * ANC >1,500/mcL
  * Platelets >100,000/mcL
  * Total bilirubin < or equal to 1.5 X ULN
  * AST(SGOT)/ALT(SGPT) < or equal to 2.5 X ULN OR < or equal to 5.0 X ULN if considered due to tumor
  * Amylase/Lipase < or equal to 1.5 X ULN
  * Alkaline Phosphatase < or equal to 2.5 X ULN or </= 5 X ULN if considered tumor related.
  * Potassium, magnesium, calcium, phosphorus, creatinine WNL prior to randomization
  * OR
  * Creatinine clearance of > 50 calculated by cockroft-gault formula
* WOCBP must have negative pregnancy test within 7 days of first treatment and use appropriate contraception.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Have received nilotinib or additional tyrosine kinase inhibitors or additional targeted therapies (except for imatinib).
* May not be receiving any other investigational agents within 4 weeks before treatment.
* Prior or concomitant malignancies (with a relapse in the last 5 years or requiring active treatment) other than GIST and with exception of previous or concomitant basal cell skin, previous cervical carcinoma in situ.
* Impaired cardiac function, including any one of the following:

Complete left bundle branch block. Ventricular paced cardiac pacemaker. Congenital long QT syndrome or family history of long QT syndrome. History of or presence of symptomatic ventricular or atrial tachyarrhythmias. Clinically significant resting bradycardia (< 50 beats per minute). QTc > 480 msec on screening ECG (using the QTcF formula). If QTc > 480 msec and electrolytes are not within normal ranges (electrolytes should be corrected and then the patient rescreened for QTc).

Right bundle branch block plus left anterior hemiblock, bifascicular block. Myocardial infarction within 12 months prior to Visit 1. Other clinically significant heart diseases (e.g., unstable angina, congestive heart failure or uncontrolled hypertension).

Severe and/or uncontrolled concurrent medical disease that could cause unacceptable safety risks or compromise compliance with protocol e.g. impairment of GI function, or GI disease that may significantly alter absorption of study drugs; uncontrolled diabetes; active infections; psychiatric illness/social situation that would limit compliance with study requirements.

* Inability to remain laying down in PET scanner for up to one hour.
* Use of any medications that prolong the QT interval and CYP3A4 inhibitors if treatment cannot be either safely discontinued or switched to a different medication prior to starting study drug administration.
* Major surgery ≤ 2 weeks prior to Visit 1 or who have not recovered from side effects of such surgery.
* Known history of noncompliance to medical regimens or inability/unwillingness to return for scheduled visits, patients who are pregnant or breast feeding, patients unwilling or unable to comply with the requirements for the protocol.
* Known chronic liver disease (i.e., chronic active, hepatitis, and cirrhosis).
* Known diagnosis of HIV, currently taking combination antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Siteman Cancer Center, Washington University School of Mediciine, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the period of February 2, 2009 through May 26, 2011, recruitment occur at oncology hospital.
Period: Overall Study
Arm/Group | Nilotinib | Nilotinib + Imatinib
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib | Nilotinib + Imatinib | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression. It will be determined for both RECIST (Response Evaluation Criteria in Solid Tumors) and CHOI criteria.
Time Frame: 6 months until death or for 5 years
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Nilotinib: Nilotinib 400 mg by mouth (PO), twice daily (BID)
- Nilotinib + Imatinib: Nilotinib 400 mg twice daily (BID) with Imatinib 400 mg daily
Arm/Group | Nilotinib | Nilotinib + Imatinib
Number analyzed (Participants) | 2 | 3
weeks | 13 (5.6) | 16 (16.3)

2. Secondary Outcome: Best Overall Response Using Response Evaluation Criteria in Solid Tumors, Choi Criteria, and Positron Emission Tomography Imaging
Time Frame: Every 8 weeks for up to 5 years
Population: Too few participants to provide meaningful analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib | Nilotinib + Imatinib
Number analyzed (Participants) | 2 | 3
Participants
  Stable Disease | 2 | 0
  Partial Response | 0 | 1
  Complete Response | 0 | 0

ADVERSE EVENTS:
Arm/Group | Nilotinib | Nilotinib + Imatinib
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib (N=2) | Nilotinib + Imatinib (N=3)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholangitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial ended early due to industry support of provision of nilotinib was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No